CLINICAL TRIAL: NCT00545597
Title: A Phase III Trial of Lorenzo's Oil in Adrenomyeloneuropathy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Upon recommendation of DSMB
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD039276 (NIH); R01FD003030 (FDA)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2007-10

CONDITIONS: Adrenomyeloneuropathy; Adrenoleukodystrophy
Keywords: adrenoleukodystrophy; adrenomyeloneuropathy
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Lorenzo's oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lorenzo's oil — 4:1 glyceryl trioleate-glyceryl trierucate (Lorenzo's oil)given orally, daily as approximately 10% of nutritional calories with supplementation.

SUMMARY:
Study of the use of Lorenzo's oil in adults with adrenomyeloneuropathy, the adult form of Lorenzo's oil.

DETAILED DESCRIPTION:
This is a double-masked placebo controlled study of glyceryl trioleate-glyceryl trierucate (Lorenzo's Oil (LO)) therapy in adrenomyeloneuropathy (AMN), the adult form of X-linked adrenoleukodystrophy (X-ALD). AMN is a slowly progressive distal axonopathy that involves the long tracts of the spinal cord and differs from the rapidly progressive inflammatory cerebral forms that most commonly affect boys and adolescents. All forms of X-ALD are associated with the abnormal accumulation of very long chain fatty acids (VLCFA) in plasma and tissues. The oral administration of LO normalizes plasma VLCFA levels within 4 weeks. While previous therapeutic trials of LO therapy in patients with the cerebral forms of X-ALD have been disappointing, recent studies suggest that it is beneficial in two types of X-ALD: 1) as a preventive of neurological involvement in asymptomatic boys; and 2) in AMN, where it appears to slow the rate of progression. None of the previous studies have been controlled, and we are now conducting the first placebo-controlled trial.

The 4-year study will include 120 men with AMN who do not have evidence of cerebral involvement, and 120 women who are heterozygous for X-ALD and have an AMN-like syndrome. The rate of progression will be compared in the LO and placebo groups using the Kurtzke EDSS score as the primary outcome and a variety of secondary outcomes.

Adrenomyeloneuropathy affects about 1 in 40,000 men and 1 in 30,000 women. It is a progressive disorder that leads to inability to walk and other severe deficits. This study will provide definitive information whether Lorenzo's Oil therapy can slow progression.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 years or older in whom the diagnosis of X-ALD has been confirmed by VLCFA assay and/or mutation analysis.
* Clinical evidence of spinal cord involvement with EDSS score between 1 and 6.5. Patients with an EDSS score of 6.5 are severely affected but have retained the capacity to walk 20 meters with the aid of a walker, crutch, or two canes.
* Either a normal brain MRI, or a type 3 pattern of MRI abnormality in which the abnormality is considered to represent the centripetal extension of the distal axonopathy.
* Adrenal function assessed by measurement of plasma ACTH and appropriate steroid replacement if adrenal insufficiency is present.

Exclusion Criteria:

* Kurtzke EDSS score of >6.5.
* Cognitive or behavioral abnormalities that impair capacity to give informed consent or carry out procedures that form part of the protocol.
* Current use, or use within 3 months, of Lorenzo's oil or other therapies that may alter the course of X-ALD. Bone marrow transplant will be a permanent exclusion criterion.
* Contraindications for MRI procedure such as subjects with paramagnetic materials in the body, such as aneurysm clips, pacemakers, intraocular metal or cochlear implants.
* Subjects who are pregnant.
* Allergies to peppermint
* Presence of non-specific conditions that may interfere with clinical assessment or participation in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical Progression of the disorder | 48 months

SECONDARY OUTCOMES:
Determine the degree to which newly developed methods to assess spinal cord function and structure in adrenomyeloneuropathy, namely quantitative sensorimotor tests and spinal cord imaging, can act as early surrogate markers of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald V Raymond, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

REFERENCES:
- See also: Adrenomyeloneuropathy (AMN) Research Study — http://www.kennedykrieger.org/kki_misc.jsp?pid=6041
- See also: United Leukodystrophy Foundation — http://www.ulf.org/
- See also: Myelin Project — http://www.myelin.org/